CLINICAL TRIAL: NCT02767700
Title: Evaluation of NGS in Combination With an Oncology Treatment Decision Support Software for Evidence-based Priorization of Individualised Treatment in Patients With Pancreatic Cancer
Brief Title: NGS and TME for Evidence-based Treatment of Pancreatic Cancer
Acronym: PePaCaKa-01
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Matthias Löhr, Professor of Gastroenterology & Herpetology, Karolinska University Hospital
Other Study IDs: PePaCaKa-01
Record Dates: First submitted 2016-03-08; First posted 2016-05-10 (Estimated); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study will make use of routinely taken samples (surgical resection, biopsy)
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: NGS — Next generation sequencing

SUMMARY:
The tumor tissue of patients with pancreatic cancer will be submitted to next-generation sequencing (NGS) and these data will be evaluated with an oncology treatment decision support (TDS) software tool that is a medicinal product class 1 (CE-marked). This software will make evidence-based suggestions for drugs likely to be effective, ineffective, or toxic (FDA approved biomarkers). For patients fit for second-line therapy, the resulting recommendations will be judged by the tumor board.

DETAILED DESCRIPTION:
Tumor tissue of patients (surgical resection, biopsy) will be used for SWEDAC-certified DNA extraction and NGS. Pseudonymised sequencing data will be fed into a TDS software tool (TreatmentMAP™, Molecular Health) and based on published evidence, suggestions will be made, graded into NCCN categories of approved drugs in indication or otherwise, clinical evidence or experimental. Same with anticipated inefficacy. In addition, FDA-approved biomarkers for toxicity will be analysed. This information is taken to the tumor board for making a decision whether this information is useful and eventually to recommend a treatment for a given patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 years up to 75 years
* Patient willing and able to provide informed consent
* TreatmentMAP™ NGS/TME is ordered by the tumor board (MDT) under routine clinical practice
* Diagnosis of a locally advanced, inoperable or metastatic pancreatic carcinoma, clinically and histologically verified according to the currently prevailing standards.
* Patient received first line therapy according to applicable guidelines and/or standards (SoC)
* Sufficient testing material available (e.g. tumor biopsy) to allow NGS/TME NGS panel testing.

Exclusion Criteria:

* Patients with ongoing systemic infection,
* Patients with immunodeficiency,
* Patients with severe cardiovascular and pulmonary morbidity that might interfere with or preclude further systemic anticancer treatment,
* Patients on full therapeutic anticoagulation.
* Patients who, due to their clinical status, are not eligible for further systemic anticancer therapy (chemotherapy, immunotherapy etc.)
* Patients who, due to their disease status are in need of immediate therapy and cannot wait for the result of the NGS/TME process.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic adenocarcinoma
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2016-04; Primary Completion 2018-03-25 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with technical success | 2 weeks

SECONDARY OUTCOMES:
Number of participants with actionable targets | 3 days
  actionable targets (effective, ineffective, FDA approved toxicity markers)

OTHER OUTCOMES:
Number of patients where NGS+TME generated information was used for treatment | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Johan Permert, MD PhD, Study Chair — Karolinska University Hospital

IPD SHARING:
Plan to Share IPD: Yes
Sequencing data will be made available anonymously

REFERENCES:
- [Background] Malgerud L, Lindberg J, Wirta V, Gustafsson-Liljefors M, Karimi M, Moro CF, Stecker K, Picker A, Huelsewig C, Stein M, Bohnert R, Del Chiaro M, Haas SL, Heuchel RL, Permert J, Maeurer MJ, Brock S, Verbeke CS, Engstrand L, Jackson DB, Gronberg H, Lohr JM. Bioinformatory-assisted analysis of next-generation sequencing data for precision medicine in pancreatic cancer. Mol Oncol. 2017 Oct;11(10):1413-1429. doi: 10.1002/1878-0261.12108. Epub 2017 Aug 8. PMID 28675654